CLINICAL TRIAL: NCT03885752
Title: The Effects of Preoperatively Chewing Gum on Sore Throat After General Anaesthesia With a Laryngeal Mask
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Tingting Wang, Director, Principal Investigator, Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TI3WT
Record Dates: First submitted 2019-03-17; First posted 2019-03-22 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Postoperative Sore Throat

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (Active Comparator)
  Interventions: Other: swallow twice
- the gum group (Placebo Comparator)
  Interventions: Drug: chewed mint gum

INTERVENTIONS:
Drug: chewed mint gum — In the preoperative waiting area before transferring to the operating room, patients in group G chewed mint gum for 2 minutes and then spit it out.
  Arms: the gum group
Other: swallow twice — asked to swallow twice without any additional treatment.
  Arms: the control group

SUMMARY:
Postoperative sore throat (POST) is an important problem after general anaesthesia. We assessed whether chewing gum preoperatively can reduce the incidence of POST after general anaesthesia administered via a streamlined liner of the pharyngeal airway (SLIPA).

ELIGIBILITY:
Inclusion Criteria:

American Society of Anaesthesiologists (ASA) class I or II 20-65 years body mass index (BMI) scores <30 undergoing elective hysteroscopic surgery -

Exclusion Criteria:

chronic laryngitis chronic bronchitis asthma gastroesophageal reflux allergies to study drugs recent use of non-steroidal anti-inflammatory drugs (NSAIDs) a history of upper respiratory tract infection in the past one week Mallampati grade>2 a history of steroid therapy.

-

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of POST scores > 3 | within 24 hours after surgery
  POST was evaluated by the Numerical Rating Scale (NRS), which ranges from 0 to 10 points, with 0 indicating completely painless, 1~ 3 indicating mild discomfort, 4 ~ 6 indicating moderate pain, and 7~ 10 indicating severe pain.

SECONDARY OUTCOMES:
the POST scores | 2 hours, 6 hours and 24 hours after surgery.
  POST was evaluated by the Numerical Rating Scale (NRS), which ranges from 0 to 10 points, with 0 indicating completely painless, 1~ 3 indicating mild discomfort, 4 ~ 6 indicating moderate pain, and 7~ 10 indicating severe pain.

OTHER OUTCOMES:
subgroup analysis with patient subdivided based on whether the laryngeal mask had blood on it. | Immediately after removal of laryngeal mask
  blood stain

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of The Obstetrics and Gynecology Hospital, Fudan University,, Shanghai, China

REFERENCES:
- [Derived] Wang T, Wang Q, Zhou H, Huang S. Effects of Preoperative Gum Chewing on Sore Throat After General Anesthesia With a Supraglottic Airway Device: A Randomized Controlled Trial. Anesth Analg. 2020 Dec;131(6):1864-1871. doi: 10.1213/ANE.0000000000004664. PMID 31990730